CLINICAL TRIAL: NCT02008643
Title: Health Related Quality of Life in Children With Food Allergy: Comparison to Healthy Children and Children With Other Chronic Diseases
Brief Title: Health Related Quality of Life in Children With Food Allergy: Comparison to Controls and Other Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 12-AOI-07
Record Dates: First submitted 2013-12-03; First posted 2013-12-11 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-03

CONDITIONS: Children With Food Allergy
Keywords: Health related quality of life, food allergy, children, chronic diseases
MeSH Terms: conditions — Food Hypersensitivity; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- children with food allergy (Experimental): Chidren aged 8-18 year with food allergy
  Interventions: Other: filling questionnary to quality of life
- children with chronic diseases (Active Comparator)
  Interventions: Other: filling questionnary to quality of life
- witnesses (Active Comparator): Inclusion criteria Age between 8-18 year old Children attending schools of Nice City Signed informed consent of the two parents Signed informed consent of the child Health insurance recipient
  Non inclusion criteria Association with another medical or psychiatric chronic disease No signed consent
  Interventions: Other: filling questionnary to quality of life

INTERVENTIONS:
Other: filling questionnary to quality of life — filling questionnary to quality of life

SUMMARY:
The number of studies concerning health related quality of life (HRQL) in children with food allergy is very limited.

Only one study to date has compared HRQL of a group of children with food allergy to data published on general population and other chronic diseases. This study concluded to lowest HRQL scores in food allergic children compared to type 1 diabetes mellitus with important impact on scores concerning social activities.

DETAILED DESCRIPTION:
Primary aim:

To compare generic HRQL score in children with food allergy with other chronic diseases and with healthy chidren in an homogeneous socio-cultural context.

Secondary aims :

* To compare generic and specific HRQL scores in children with food allergy
* Identifify in chidren with food allergy, clinical factrors assocated with lowest scores in order to improve our management.

Methods

Generic HRQL questionnaire (CHQ-87) will be distributed :

* after hospital consultation for patients
* in schools for healthy children A specific HRQL questionnaire (FAQLQ-CF or TF) and the " Food Allergy Independent Measure " will also distributed to chidren with food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8-18 year old
* IgE mediated food allergy diagnosed by a pediatric allergologist with following criteria:

Convincing history of allergic reaction with positive prick-test and specific IgE Or Open food challenge associated with positive prick-test and specific IgE

* Signed informed consent of the two parents
* Signed informed consent of the child
* Health insurance recipient

Exclusion Criteria:

* Association with another medical or psychiatric chronic disease (excepted for controlled asthma)
* Partially or not controlled asthma during last year
* No signed consent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 861 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
comparison of12 scores of the generic health-related quality of life questionnaire CHQ-CF 87 between children with food allergy and healthy children scores. | Once at inclusion
  12 scores concerning the 12 following dimensions:
  * physical functioning
  * role functioning emotional
  * role functioning behavior
  * role functioning physical
  * bodily pain
  * general behavior
  * mental health
  * self-esteem
  * general health
  * change in health
  * family activities
  * family cohesion
  Comparison between children with food allergy and healthy children scores.

SECONDARY OUTCOMES:
comparaison beetween all questionnary | once at inclusion
  1. Comparison of the CHQ-CF 87 scores between children with food allergy and chidren with other chronic diseases.
  2. Comparison of the CHQ-CF 87 scores with the FAQLQ-CF (or -TF) score (global and 4 dimensions) and with the FAIM score.
  3. Comparison of the FAQLQ-CF (or-TF) (global and 4 dimensions) with clinical characteristics of the children with food allergy

CONTACTS AND LOCATIONS:
Overall Officials: Lisa GIOVANNINI-CHAMI, PH, Principal Investigator — CHU de Nice-Lenval
Locations (1):
- Service de Pédiatrie, Nice, Nice, France